CLINICAL TRIAL: NCT07154628
Title: Effect of Topical Lidocaine Spraying on the Vocal Cords Before Intubation During Robotic Surgery: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20250221
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Lidocaine Spray; Intubation; Robotic Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Active Comparator): The group of patient will receive lidocaine spraying on vocal cord before intubation
  Interventions: Drug: Normal Saline (0.9% NaCl)
- Control group (Placebo Comparator): The group of patient will receive normal saline spraying on vocal cord before intubation
  Interventions: Drug: Lidocaine %2 ampoule

INTERVENTIONS:
Drug: Lidocaine %2 ampoule — During general anesthesia, the anesthesiologist administers 1.5cc of lidocaine spraying on the vocal cords using Terumo SurfloTM I.V. Catheter 20G before intubation.
  Arms: Control group
Drug: Normal Saline (0.9% NaCl) — During general anesthesia, the anesthesiologist administers 1.5cc of normal saline spraying on the vocal cords using Terumo SurfloTM I.V. Catheter 20G before intubation.
  Arms: Lidocaine group

SUMMARY:
Endotracheal intubation is a respiratory management technique used during general anesthesia. It is essential for certain surgical procedures as it ensures a secure airway for the patient.

However, during the placement of the endotracheal tube, the passage of the tube through the vocal cords can cause pain stimulation, leading to an increase in heart rate and blood pressure. Lidocaine reversibly blocks the conduction of nerve impulses along nerve fibers by preventing the movement of sodium ions across the nerve membrane. Topical application of lidocaine near the vocal cords before endotracheal tube placement may be a way to reduce the surgical pleth index and changes in vital signs (heart rate, blood pressure) caused by excessive endotracheal tube stimulation.

This study aims to investigate the benefit of topical spraying of lidocaine on the vocal cords before endotracheal tube placement during routine da Vinci surgery. The primary outcomes were the pharmacological effects of spraying either lidocaine or normal saline (control group) on the vocal cords. These included: post-intubation hypertension (defined as an increase in systolic blood pressure of more than 20% from baseline), changes in mean arterial pressure before and after intubation, and objective pain indices such as the Surgical Pleth Index. Secondary outcomes included post-intubation hypotension (defined as mean arterial pressure less than 70 mmHg), as well as postoperative complaints and severity of sore throat, pain on swallowing, and hoarseness.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I~III
* aged 18~69 y/o
* BMI 18~35 kg/m2
* scheduled for elective robotic surgery under general anesthesia

Exclusion Criteria:

* Allergy or contraindication to lidocaine

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
post-intubation hypertension | From enrollment to the end of surgery
  defined as an increase in systolic blood pressure of more than 20% from baseline
changes in mean arterial pressure before and after intubation | From enrollment to the end of surgery
objective pain indices (Surgical Pleth Index) | From enrollment to the end of surgery

SECONDARY OUTCOMES:
post-intubation hypotension | From enrollment to postoperative day 1
  defined as mean arterial pressure less than 70 mmHg
postoperative sore throat | From enrollment to postoperative day 1
  During patients' stay in post-anesthetic care unit and our postoperative follow-up visiting at postoperative day 1, we will check the patients if they have any complaint of postoperative sore throat.
pain on swallowing | From enrollment to postoperative day 1
  During patients' stay in post-anesthetic care unit and our postoperative follow-up visiting at postoperative day 1, we will check the patients if they have any complaint of pain on swallowing.
hoarseness | From enrollment to postoperative day 1
  During patients' stay in post-anesthetic care unit and our postoperative follow-up visiting at postoperative day 1, we will check the patients if they have any complaint of hoarseness.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
New analyses often require additional ethics committee approval.